CLINICAL TRIAL: NCT04261452
Title: Heart Failure Worsens Leg Muscle Strength and Endurance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Heart Failure Worsens Muscle Strength in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayron Faria de Oliveira (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Sponsor-Investigator, Mayron Faria de Oliveira, Clinical Investigator, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 1275295
Record Dates: First submitted 2020-02-03; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: COPD; CHF; Muscle Weakness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscle Weakness | interventions — Exercise Test; Respiratory Function Tests; Echocardiography, Doppler; Anthropometry; Body Composition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPD (Other): Body composition was assessed using a body composition. The same medical doctor performed all echocardiograms and all patients underwent comprehensive M-mode echocardiography. Spirometry, gas transfer and static lung volumes were measured in all patients. Resting blood gases were obtained by samples from the radial artery. The six-minute walk test and the four-minute step test were performed. All CPET tests were performed on an electronically braked cycle ergometer and standard metabolic and ventilatory responses were measured breath-by-breath using a calibrated, computer-based system. Knee flexors and extensors muscles were analysed by an isokinetic dynamometer. All patients performed two maximal isokinetic tests: 6 repetitions at 60°/s and 20 repetitions at 300°/s.
  Interventions: Diagnostic Test: isokinetic dynamometer; Diagnostic Test: Cardiopulmonary Exercise Test; Diagnostic Test: Functional Capacity Tests; Diagnostic Test: Lung Function Test; Diagnostic Test: Doppler Echocardiography; Diagnostic Test: Anthropometry and Body Composition
- Overlap (Other): Body composition was assessed using a body composition. The same medical doctor performed all echocardiograms and all patients underwent comprehensive M-mode echocardiography. Spirometry, gas transfer and static lung volumes were measured in all patients. Resting blood gases were obtained by samples from the radial artery. The six-minute walk test and the four-minute step test were performed. All CPET tests were performed on an electronically braked cycle ergometer and standard metabolic and ventilatory responses were measured breath-by-breath using a calibrated, computer-based system. Knee flexors and extensors muscles were analysed by an isokinetic dynamometer. All patients performed two maximal isokinetic tests: 6 repetitions at 60°/s and 20 repetitions at 300°/s.
  Interventions: Diagnostic Test: isokinetic dynamometer; Diagnostic Test: Cardiopulmonary Exercise Test; Diagnostic Test: Functional Capacity Tests; Diagnostic Test: Lung Function Test; Diagnostic Test: Doppler Echocardiography; Diagnostic Test: Anthropometry and Body Composition

INTERVENTIONS:
Diagnostic Test: isokinetic dynamometer — Knee flexors and extensors muscles were analysed by an isokinetic dynamometer. Positioning of the subjects (sitting with hips flexed to 75°) was standardized based on the length of the thigh and leg to minimize individual differences. Correction for the effect of gravity on neuromuscular performance was accomplished by incorporating limb mass into the calculation of torque production. Previous warm-up was repeated five time with an angular velocity of 400°/s. All patients randomly performed two maximal isokinetic tests: 6 repetitions at 60°/s and 20 repetitions at 300°/s.
  Measurements of torque, work (J), power (W) maximum (peak), and fatigue index were obtained in both tests. In addition, data were analysed at percent of prediction (percent pred) by reference values previously described for the Brazilian population, corrected by muscle mass and peak values.
  Other Names: Muscle Performance
Diagnostic Test: Cardiopulmonary Exercise Test — All exercise tests were performed on an electronically braked cycle ergometer. Standard metabolic and ventilatory responses were measured breath-by-breath using a calibrated, computer-based system.
  The incremental exercise test started with 2-min unloaded cycling and increments of 3-10 Watts per min until exhaustion. The anaerobic threshold was estimated by the ventilatory equivalents and V-slope methods and it was determined in agreement by a cardiologist and pulmonologist. Heart rate was determined using the 12-lead electrocardiogram. Throughout the experiment, the pulse hemoglobin saturation (SpO2) was assessed with a pulse oximeter and the 'shortness of breath' was asked at exercise cessation using the 0-10 Borg category ratio scale. All measurements were expressed as percentage predicted for the Brazilian population.
Diagnostic Test: Functional Capacity Tests — The six-minute walk test (6MWT) was in accordance with the American Thoracic Society (ATS). The four-minute step test (4MST) consisted of going up and down a 20-cm high, 40-cm wide and 40-cm long step for 4 minutes.
  The investigators measured the heart rate and pulse hemoglobin saturation at rest before each test and every minute of both tests. The investigators assessed dyspnoea and leg fatigue at rest and with the modified Borg scale immediately after finishing the test.
Diagnostic Test: Lung Function Test — Spirometry, gas transfer, and static lung volumes were measured in all patients, and airflow was measured using a "Pitot-tube" based on the American Thoracic Society/European Respiratory Society guidelines. Measurement of maximal inspiratory and expiratory pressures was performed from the residual volume and total lung capacity. Resting blood gases were obtained by samples from the radial artery.
Diagnostic Test: Doppler Echocardiography — The same medical doctor performed all echocardiograms and all patients underwent comprehensive echocardiography.
Diagnostic Test: Anthropometry and Body Composition — Body composition was assessed using a body composition analyzer. Percent body fat was estimated from the resistance and reactance values.
  Resistance values and the subject's height (meters), weight (kg), sex, and age (years) were entered into a computer program to estimate percentage of fat, fat mass (FM), and muscle mass (MM).

SUMMARY:
The combination of heart failure (HF) and chronic obstructive pulmonary disease (COPD) is highly prevalent, but underdiagnosed and poorly recognized. It has been suggested that the decline in functional capacity is associated with musculoskeletal and systemic changes than primary organ (heart and/or lung) failure. In addition, it is recognized that both diseases have several mechanisms that are responsible for musculoskeletal impairment. However, the association of reduced systemic perfusion with low oxygen content observed in the association of HF and COPD may contribute to the worsening of the components of the muscle impairment cascade. Thus, muscle strength and fatigue may not only be even more altered but may also be the main determinants of functional capacity in patients with coexistence of HF and COPD. Although many studies have evaluated the muscle performance of patients with HF or COPD, the literature did not show data on worsening due to the association of the diseases. Particularities identification of the muscle impairment in the coexistence of HF and COPD is fundamental for the development of rehabilitation strategies, mainly through physical exercise. In this line, the present study tested the hypothesis that the coexistence of HF and COPD could present lower values of strength and greater fatigue. Similarly, the muscle dysfunction degree could strongly correlate with the performance markers of the incremental or functional tests in patients with HF associated with COPD.

The study protocol was reviewed and approved by the Institutional Research Board. All subjects gave written informed consent before participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* non-cachectic sedentary patients
* moderate-to-severe COPD according to GOLD classification (FEV1/ FVC <0.7 and predicted post-bronchodilator FEV1 between 30% and 80%)
* no clinical or echocardiographic evidence of HF for the COPD group
* echocardiographic evidence of HF with reduced left ventricular ejection fraction (<40%) for the overlap group
* chronic dyspnoea (MRC scale score 2-4)
* NYHA class 2 or 3.

Exclusion Criteria:

* long-term O2 therapy
* recent (within a year) rehabilitation program
* osteomuscular limitation
* type I or non-controlled type II diabetes mellitus
* peripheral arterial disease associated with claudication
* Patients with preserved ejection fraction HF

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Muscle weakness | one week after all tests
  Muscle performance will be assessed by an isokinetic dynamometer. All data will be measured in absolute values and the percentage of predicted values for the Brazilian population.
Cardiopulmonary function | one week after all tests
  Exercise capacity will be assessed by the cardiopulmonary test. All data will be measured in absolute values (ml/kg) and the percentage of predicted values for the Brazilian population.
Clinical tests | one day after all tests
  Performance in clinical tests will be assessed by 6MWT and 4-min Step test. All data will be measured in absolute values.
Lung Function | one day after all tests
  Clinical obstruction data will be assessed by total body plethysmography. All data will be measured in absolute values and percentage of predicted values for the Brazilian population.
Cardiac Function | one day after all tests
  An echocardiogram will be performed to assess all cardiac functions. All data will be measured in the percentage of predicted values for the Brazilian population.
Body composition | one day after all tests
  Fat-free mass will be assessed by body composition. All data will be measured in the percentage of predicted values for the Brazilian population.

IPD SHARING:
Plan to Share IPD: No